CLINICAL TRIAL: NCT05791721
Title: Preemptive Use of Etoricoxib and Dexamethasone: Effect on Early Bone Healing, Inflammatory Response, and Postoperative Parameters After Impacted Lower Third Molar Surgery
Brief Title: Effect of Preemptive Etoricoxib and Dexamethasone on Wound Healing and Clinical Parameters After Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Iva Mijailovic, Principal Investigator, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 36/22
Record Dates: First submitted 2023-03-04; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Surgical Wound; Post Operative Pain
Keywords: Third Molar; Analgesia; Saliva
MeSH Terms: conditions — Surgical Wound; Pain, Postoperative; Agnosia | interventions — Etoricoxib; Tablets; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Etoricoxib group (Active Comparator): One hour preoperatively, preemptive, single-dose etoricoxib tablet in dosage of 90 mg will be administered orally
  Interventions: Drug: Etoricoxib 90 Mg Oral Tablet
- Dexamethasone group (Active Comparator): One hour preoperatively, preemptive, single-dose dexamethasone in dosage of 4 mg will be administered intramuscularly
  Interventions: Drug: Dexamethasone 4mg
- Control group (No Intervention): In this group, one hour preoperatively no medication will be administered

INTERVENTIONS:
Drug: Etoricoxib 90 Mg Oral Tablet — Intervention will be applied one hour before surgical extraction of impacted mandibular third molar
  Other Names: There is no other intervention name
  Arms: Etoricoxib group
Drug: Dexamethasone 4mg — Intervention will be applied one hour before surgical extraction of impacted mandibular third molar
  Other Names: There is no other intervention name
  Arms: Dexamethasone group

SUMMARY:
The goal of this clinical trial is to compare preemptive single-dose selective cyclooxygenase 2 (COX-2) inhibitor - etoricoxib and dexamethasone use in systemically healthy patients during the surgical extraction of impacted mandibular third molars. The main questions it aims to answer/evaluate are:

* the level of inflammatory and early wound healing mediators in patients' saliva during early postoperative phase
* clinical postoperative parameters such as pain, swelling and trismus
* patient satisfaction with the treatment
* rescue medication consumed during the postoperative period
* incidence of adverse events

Participants indicated for mandibular third molar surgery will be asked to:

* take premedication (etoricoxib or dexamethasone) before surgical extraction
* provide saliva samples before and following the surgery at regular check-ups
* note the amount of rescue medication taken and pain intensity in different time points
* perform clinical measurements of swelling and trismus at regular check-up visits
* answer the questions about satisfaction and potential adverse events, if occur Researchers will compare preemptive single-dose etoricoxib, preemptive single-dose dexamethasone, and no premedication in impacted mandibular third molar surgery, to see if there are differences in inflammatory response and early wound healing, as well as in clinical postoperative parameters, patient satisfaction with the treatment and incidence of potential adverse events.

DETAILED DESCRIPTION:
Acute pain, swelling and trismus present typical clinical manifestation following impacted mandibular third molar surgery. Postoperative wound healing is regulated by activity of inflammatory mediators and osteogenic factors. Nonsteroidal anti-inflammatory drugs, especially cyclooxygenase 2 (COX-2) inhibitors and glucocorticoids are routinely used to improve postoperative clinical state of the patients. Studies have shown that both COX-2 inhibitors and dexamethasone may decrease the number of postsurgical rescue medication intake, reduce the postoperative edema and increase the mouth opening ability. Analgesic efficacy of etoricoxib (ETOX), a high selective COX-2 inhibitor has been shown as superior compared to placebo and other nonsteroidal anti-inflammatory drugs in third molar surgery. However, literature data on comparative testing of ETOX and dexamethasone (DEX) use in third molar surgery are scarce. Furthermore, no studies with a 7 days follow-up were conducted. Preclinical studies indicate that COX-2 inhibitors and DEX may negatively affect early wound healing by down-regulation of mediators such as COX-2, prostaglandin E2 (PGE2), alkaline phosphatase (ALP), runt-related transcription factor 2 (RUNX2), and osteocalcin (OCN). Specialized pro-resolving lipid mediators are important for resolution phase of inflammatory process and wound healing. According to animal studies, maresin 1 (MAR1) has important role in post-trauma pain reduction and bone healing, thus the expression of this mediator may be significant to indicate the course of postoperative wound healing. In the current literature, no data on salivary early bone healing mediators following preemptive use of ETOX and DEX in mandibular third molar removal are available. Moreover, the correlation of these markers, as well as inflammatory saliva mediators with the clinical parameters may be important for potential developing of future unique protocols for premedication in third molar surgery.

The primary goal of the research will be to evaluate the level of inflammatory and early wound healing mediators (COX-2, PGE2, ALP, RUNX2, OCN, MAR1) in saliva samples obtained from the systemically healthy patients requiring impacted mandibular third molar extraction, in conditions of 1-preemptive single-dose ETOX 90 mg oral use; 2-preemptive single-dose DEX 4 mg intramuscular use, and 3-no premedication. Secondary outcomes will include correlation of mentioned salivary mediators with postoperative clinical parameters such as pain, swelling and trismus. Furthermore, rescue medication intake, patient satisfaction with the treatment, and incidence of potential adverse events will be recorded.

A prospective, randomized, controlled, parallel-group, double-blinded clinical trial will be conducted at the Department of Oral surgery and Laboratory for basic science, School of Dental medicine, University of Belgrade, Serbia. The research will be performed following the CONSORT guidelines, per the Helsinki Declaration. Subjects who require unilateral fully impacted mandibular third molar extraction will be screened for eligibility. After meeting the inclusion criteria, participants will receive verbal and written information on the study objectives, protocol as well as the possible risks and benefits of the study. Only the eligible subjects who agree with the information provided and sign an informed consent form will be enrolled in the study. A total of 90 patients will be included (n=30). Computer-generated blocked randomization with a 1:1:1 allocation ratio (block size 6) will be performed by a researcher not included in the study (Microsoft Excel, version 2016). To conceal the allocation, the papers containing a code of the allocated group (1-ETOX group; 2-DEX group; 3-control group) will be sequentially packed in opaque envelopes and sealed. One hour before the intervention, the same independent researcher will unseal the following envelope and, depending on the study group, administer ETOX in a blurred plastic container (ETOX group), DEX in the unspecified syringe (DEX group), or provide written information on cold packs usage during the postoperative period (control group). The patients will be unaware of the generic and the brand name of the medications, but they will be notified that the drugs are registered and on the market. The allocation will be concealed until the finishing of the data analysis. The surgeon who will perform all the interventions and the researcher who will collect the data will be masked to the patients' allocations.

After recruitment, data on age (years), sex, and smoking status (no smoking, ≤10/day, or >10/day) will be obtained from all the included patients. During the same visit, the surgical intervention will be scheduled, and the third molar position will be estimated on panoramic radiographs, according to the Pell and Gregory and Winter classifications. Initial exam, pre-, perioperative, and follow-up measurements will be performed by one blinded clinician.

On the second study visit, one hour before surgical intervention, patients will be instructed to note the amount of pain experienced at that moment on a 10-cm long visual analog scale (VAS), where 0 means no pain at all and 10 represent the greatest pain they ever felt. A 6-point verbal rating pain scale (VRS) will be also provided to the patients to document the current pain (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain). Additionally, baseline measurements of a maximal inter-incisor and lobule-pogonion distance at the side of the extraction-required third molar in millimeters will be obtained by a soft tape measure. Afterward, 1 hour before the surgery patients will receive: single-dose ETOX 90 mg (Etoxib®, KRKA, Novo Mesto, Slovenia) orally (ETOX group); single-dose DEX 4 mg (Dexason®, Galenika, Belgrade, Serbia) in deltoid muscle (DEX group); no premedication (control group).

After regional inferior alveolar, lingual, and buccal nerve blocks with a local anesthetic consisting of 4% articaine hydrochloride with 1:100000 epinephrine (Septanest®, Septodont, Saint-Maur-des-Fosses, France), the surgical removal of impacted mandibular third molar will be performed according to the technique previously described in the literature: after full-thickness flap elevation, bone removal will be performed by rotatory instruments under sterile saline irrigation. Instruments such as levers will be used for tooth extraction, and tooth separation will be performed, if necessary. After tooth extraction and bone edges smoothening, the wound will be primary sutured. All the surgical procedures will be performed by one experienced oral surgeon, masked to the allocation group. Perioperatively, the duration of the intervention (min), the amount of local anesthetic solution used (ml), tooth separation if performed, and any complications such as inferior alveolar vascular damage will be registered.

Following the intervention, patients will be advised to take rescue medication if pain occurs at any time. Paracetamol 500 mg regimen will be prescribed as an escape analgesic (Paracetamol®, Galenika, Belgrade, Serbia), with the instructions to not exceed the maximal recommended daily dose (4000 mg). Additionally, the antibiotics will be prescribed: amoxicillin 500 mg or clindamycin 600 mg in case of penicillin hypersensitivity, three times a day for 5 days. Thereafter, all the patients will receive written hygienic-dietary instructions with the advice of careful oral hygiene maintenance, a soft diet, avoidance of mouth rinsing, as well as smoking, hot food, and hot beverages. The additional penned information for the control group will involve repeated use of cold packs with a 20-min pause, and will be submitted to the patients preoperatively.

After surgery, patients will received a pre-designed take-home diary containing fields for rescue analgesic registration (every time of intake, number of the regimen, and dose) and a list of the most common adverse events (headache, nausea, vomiting, vertigo, insomnia, fever), with instructions to check any of the listed, or write down any other if occurred. Additionally, patients will be instructed to record pain intensity on VAS and VRS at 2h, 4h, 6h, 8h, 10h, 12h, and 72h following the surgery, as well as in every case of rescue medication intake.

Control check-ups will be scheduled at 24h, 48h, and 7 days postoperatively. On each control examination, the 5-point Likert scale will be used to assess patient satisfaction at the respective time. The following question will be asked: "How satisfied are you at this moment with the impacted mandibular third molar surgery?", and the possible answers will be: "5-very satisfied", "4-satisfied", "3-neutral", "2-dissatisfied", and "1-very dissatisfied". After collecting the answers from every check-up visit, average patient satisfaction with the treatment will be calculated. During every control study visit, the severity of pain experiencing at that moment will be noted on VAS and VRS. Maximal inter-incisor and lobule-pogonion distance on the operated side will be measured. In addition, at a 7-day check-up the take-home diary will obtained from the patients.

Samples containing 0,5 ml of unstimulated saliva will be collected from the floor of the mouth by means of 2 ml plastic syringe and dull needle of 18 Gauge thickness in four time points: One hour before surgery, immediately, 48h and 7 days after the surgery. Saliva samples will be collected in sterile plastic tubes that are pre-filled with fluid that prevents RNA degradation and stored at -80 degrees Celsius until laboratory analysis.

Laboratory procedures will be performed with aim to assess the level of relative gene as well as protein expression of inflammatory (COX-2, PGE2) and early wound healing (RUNX2, ALP, OCN, MAR1) mediators in tested groups in different time points of interest. After RNA isolation and obtaining of complementary DNA (according to the manufacturer instructions), relative gene expression of COX-2, PGE2, RUNX2, ALP and OCN will be evaluated by means of real-time polymerase chain reaction assay. Protein expression of PGE2 and MAR1 will be performed by enzyme linked immunosorbent assay (ELISA).

Statistical analysis will be performed in statistical package SPSS, version 22.0 (SPSS, Inc. Chicago). Data will be presented through mean, standard deviation, median, maximum and minimum values, percent. Depending of the data distribution, appropriate parametric or non-parametric tests will be performed. Regression models will be performed to determine the predictors of detected inter-group differences. The level of significance will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals (ASA I by American Society of Anesthesiologists classification);
* Age 18-30 years;
* Absence of hypersensitivity to any of the medications in the study;
* Subjects capable to understand the protocol and sign an informed consent form.

Exclusion Criteria:

* Systemic disorders;
* Individuals in gestation or lactation period;
* Radiographic presence of potential cystic or tumorous lesions in the region of the extraction-required IMTM;
* Any symptoms or clinical signs of the infection caused by the extraction-required IMTM up to 10 days preoperatively;
* Use of NSAIDs or corticosteroids within 10 days before the surgery.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-12-26 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
Relative gene expression of inflammatory and early wound healing salivary mediators during impacted mandibular third molar surgery in conditions of preemptive etoricoxib, dexamethasone, or no premedication use | 1 hour before surgery
  To measure the relative gene expression of COX-2, PGE2, ALP, RUNX2, OCN in saliva samples obtained 1 hour before surgical removal of impacted mandibular third molar
Protein expression of inflammatory and early wound healing salivary mediators during impacted mandibular third molar surgery in conditions of preemptive etoricoxib, dexamethasone, or no premedication use | 1 hour before surgery
  To measure the protein expression of PGE2 and MAR1 in saliva samples obtained 1 hour before surgical removal of impacted mandibular third molar
Relative gene expression of inflammatory and early wound healing salivary mediators during impacted mandibular third molar surgery in conditions of preemptive etoricoxib, dexamethasone, or no premedication use | immediately after surgery
  To measure the relative gene expression of COX-2, PGE2, ALP, RUNX2, OCN in saliva samples obtained immediately after surgical removal of impacted mandibular third molar
Protein expression of inflammatory and early wound healing salivary mediators during impacted mandibular third molar surgery in conditions of preemptive etoricoxib, dexamethasone, or no premedication use | immediately after surgery
  To measure the protein expression of PGE2 and MAR1 in saliva samples obtained immediately after surgical removal of impacted mandibular third molar
Relative gene expression of inflammatory and early wound healing salivary mediators during impacted mandibular third molar surgery in conditions of preemptive etoricoxib, dexamethasone, or no premedication use | 48 hours after surgery
  To measure the relative gene expression of COX-2, PGE2, ALP, RUNX2, OCN in saliva samples obtained 48 hours after surgical removal of impacted mandibular third molar
Protein expression of inflammatory and early wound healing salivary mediators during impacted mandibular third molar surgery in conditions of preemptive etoricoxib, dexamethasone, or no premedication use | 48 hours after surgery
  To measure the protein expression of PGE2 and MAR1 in saliva samples obtained 48 hours after surgical removal of impacted mandibular third molar
Relative gene expression of inflammatory and early wound healing salivary mediators during impacted mandibular third molar surgery in conditions of preemptive etoricoxib, dexamethasone, or no premedication use | Day 7 after surgery
  To measure the relative gene expression of COX-2, PGE2, ALP, RUNX2, OCN in saliva samples obtained on Day 7 after surgical removal of impacted mandibular third molar
Protein expression of inflammatory and early wound healing salivary mediators during impacted mandibular third molar surgery in conditions of preemptive etoricoxib, dexamethasone, or no premedication use | Day 7 after surgery
  To measure the protein expression of PGE2 and MAR1 in saliva samples obtained on Day 7 after surgical removal of impacted mandibular third molar

SECONDARY OUTCOMES:
Evaluation of preoperative pain on visual analog scale | 1 hour before surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 2 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 4 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 6 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 8 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 10 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 12 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 24 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 48 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Hour 72 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of postoperative pain on visual analog scale | Day 7 after surgery
  Pain will be measured on a 10-cm long visual analog scale (VAS), where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Evaluation of preoperative pain on verbal rating scale | 1 hour before surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 2 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 4 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 6 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 8 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 10 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 12 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 24 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 48 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Hour 72 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of postoperative pain on verbal rating scale | Day 7 after surgery
  Pain will be measured on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Evaluation of preoperative lobule-pogonion distance | 1 hour before surgery
  Baseline lobule-pogonion distance will be measured on the side requiring operation by means of a soft tape, and expressed in millimeters (mm).
Evaluation of postoperative swelling | Hour 24 after surgery
  Postoperative swelling will be assessed through measurement of lobule-pogonion distance on the operated side by means of a soft tape, and expressed in millimeters (mm).
Evaluation of postoperative swelling | Hour 48 after surgery
  Postoperative swelling will be assessed through measurement of lobule-pogonion distance on the operated side by means of a soft tape, and expressed in millimeters (mm).
Evaluation of postoperative swelling | Day 7 after surgery
  Postoperative swelling will be assessed through measurement of lobule-pogonion distance on the operated side by means of a soft tape, and expressed in millimeters (mm).
Evaluation of preoperative maximal inter-incisor distance | 1 hour before surgery
  Maximal inter-incisor distance at baseline will be measured by means of a soft tape, and expressed in millimeters (mm).
Evaluation of postoperative trismus | Hour 24 after surgery
  Trismus will be measured through assessment of a maximal inter-incisor distance by means of a soft tape, expressed in millimeters (mm).
Evaluation of postoperative trismus | Hour 48 after surgery
  Trismus will be measured through assessment of a maximal inter-incisor distance by means of a soft tape, expressed in millimeters (mm).
Evaluation of postoperative trismus | Day 7 after surgery
  Trismus will be measured through assessment of a maximal inter-incisor distance by means of a soft tape, expressed in millimeters (mm).
Patient satisfaction with the treatment | Hour 24 after surgery
  Patient will mark their satisfaction with the treatment using 5-point Likert scale. The question that will be asked to the patients will be as follows: "How satisfied are you at this moment with the impacted mandibular third molar surgery?". Possible answers on the 5-point Likert scale would be: "5-very satisfied", "4-satisfied", "3-neutral", "2-dissatisfied", and "1-very dissatisfied". Higher scores mean better outcome.
Patient satisfaction with the treatment | Hour 48 after surgery
  Patient will mark their satisfaction with the treatment using 5-point Likert scale. The question that will be asked to the patients will be as follows: "How satisfied are you at this moment with the impacted mandibular third molar surgery?". Possible answers on the 5-point Likert scale would be: "5-very satisfied", "4-satisfied", "3-neutral", "2-dissatisfied", and "1-very dissatisfied". Higher scores mean better outcome.
Patient satisfaction with the treatment | Day 7 after surgery
  Patient will mark their satisfaction with the treatment using 5-point Likert scale. The question that will be asked to the patients will be as follows: "How satisfied are you at this moment with the impacted mandibular third molar surgery?". Possible answers on the 5-point Likert scale would be: "5-very satisfied", "4-satisfied", "3-neutral", "2-dissatisfied", and "1-very dissatisfied". Higher scores mean better outcome.
Rescue medication intake | At any time during 7 days of follow up
  Patients will be instructed to note each rescue medication intake.
Day of rescue medication intake | At any time during 7 days of follow up
  Patients will be instructed to note the day when each rescue medication has been taken. Options provided to the patients would be: Day 0, Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7.
Time of rescue medication intake in hours | At any time during 7 days of follow up
  Patients will be instructed to note the time in hours (h) when each rescue medication has been taken.
Time of rescue medication intake in minutes | At any time during 7 days of follow up
  Patients will be instructed to note the time in minutes (min) when each rescue medication has been taken.
Pain intensity on visual analog scale during each rescue medication intake | At any time during 7 days of follow up
  Patients will be instructed to note pain intensity during each rescue medication intake on visual analog scale where 0 means no pain at all, and 10 represent the greatest pain patients have ever felt. Higher scores on a scale mean worse outcome.
Pain intensity on verbal rating scale during each rescue medication intake | At any time during 7 days of follow up
  Patients will be instructed to note pain intensity during each rescue medication intake on a 6-point verbal rating pain scale (VRS) where higher scores mean worse outcome (1-no pain; 2-mild pain; 3-moderate pain; 4-severe pain; 5-very severe pain; 6-the worst possible pain).
Dosage of each rescue medication intake | At any time during 7 days of follow up
  Patients will be instructed to note the dosage of each rescue medication used.
Incidence of adverse events | At any time during 7 days of follow up
  Patients will be instructed to write any postoperative adverse event if occurs

CONTACTS AND LOCATIONS:
Overall Officials: Aleksa B Markovic, Study Chair — School of Dental Medicine, University of Belgrade
Locations (1):
- School of Dental medicine, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available only to researcher who will enroll the participants and collect the data

REFERENCES:
- [Background] Martins-de-Barros AV, Barros AM, Siqueira AK, Lucena EE, Sette de Souza PH, Araujo FA. Is Dexamethasone superior to Ketorolac in reducing pain, swelling and trismus following mandibular third molar removal? A split mouth triple-blind randomized clinical trial. Med Oral Patol Oral Cir Bucal. 2021 Mar 1;26(2):e141-e150. doi: 10.4317/medoral.24088. PMID 33247572
- [Derived] Mijailovic I, Janjic B, Milicic B, Todorovic A, Ilic B, Misic T, Markovic N, Markovic A. Comparison of preemptive etoricoxib and dexamethasone in third molar surgery - a randomized controlled clinical trial of patient-reported and clinical outcomes. Clin Oral Investig. 2023 Sep;27(9):5263-5273. doi: 10.1007/s00784-023-05146-4. Epub 2023 Jul 14. PMID 37452140
- See also: The study was conducted with ASA I individuals who were submitted to preemptive 8mg dexamethasone or 20mg ketorolac tromethamine 1h before surgical third molar extraction — http://pubmed.ncbi.nlm.nih.gov/33247572/